CLINICAL TRIAL: NCT02515045
Title: Comparison of Dropless Prophylaxis After Routine Phacoemulsification to Standard Drops Regimen
Brief Title: Dropless vs. Standard Drops Contralateral Eye Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEP 14-002
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Cataract
Keywords: Cataract; Surgery; Prophylaxis
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin; nepafenac; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TriMoxiVanc (Active Comparator): The formulation containing triamcinolone acetonide, moxifloxacin hydrochloride and vancomycin used as an injection at the end of the uneventful phacoemulsification procedure. The compounded Tri-Moxy-Vanco will be delivered into the vitreous cavity using a transzonular approach after IOL implantation before removal of the OVD.
  Interventions: Drug: TriMoxiVanc
- TriMoxiVanc + Ilevro (Active Comparator): Nepafenac ophthalmic suspension 0.3% will be started 3 days prior to surgery QD and continue QD for 4 weeks after surgery. The compounded Tri-Moxy-Vanco will be injected into the vitreous cavity using a transzonular approach after IOL implantation before removal of the OVD.
  Interventions: Drug: TriMoxiVanc; Drug: Ilevro
- Control (Active Comparator): Moxifloxacin HCl 0.1%, 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  Nepafenac ophthalmic suspension 0.3% : 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Prednisolone acetate 1% will be started after surgery QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
  Interventions: Drug: Moxifloxacin HCl 0.5%; Drug: Ilevro; Drug: Prednisolone acetate 1%

INTERVENTIONS:
Drug: TriMoxiVanc — triamcinolone acetonide 15 mg / ml with moxifloxacin 1 mg/ml, vancomycin 10 mg/ml to be injected at time of cataract surgery.
  Other Names: Dropless
  Arms: TriMoxiVanc; TriMoxiVanc + Ilevro
Drug: Moxifloxacin HCl 0.5% — Antibiotic to be used 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  Other Names: Vigamox, Moxeza
  Arms: Control
Drug: Ilevro — NSAID to be used 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Other Names: Nepafenac 0.3%
  Arms: Control; TriMoxiVanc + Ilevro
Drug: Prednisolone acetate 1% — Steroid to be started after surgery 1 drop QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
  Other Names: Pred Forte, Econopred Plus, Omnipred
  Arms: Control

SUMMARY:
To compare the use of an injectable compound containing an antibiotic and an anti-inflammatory at time of cataract surgery to standard of care that is the use 3 different topical medications to prevent inflammation and infection after routine cataract surgery.

DETAILED DESCRIPTION:
Key factors for a successful cataract surgery include, among others, preoperative measurements for accurate intraocular lens (IOL) calculation, surgical technique and surgeon's experience but also the use of prophylactic topical antibiotics and anti-inflammatories (steroidal and non-steroidal, NSAID) to decrease the risk of postoperative infection (i.e. endophthalmitis) and intraocular inflammation (i.e. macular edema, CME).

Even though, the large body of literature that supports the significance of prophylactic eye drops prior to surgery, patient compliance is a common problem. Different factors have been associated with patient's lack of compliance. It could be due to patient's inability to self administer the drops, lack of understanding of the importance of using the prophylactic treatment as well as understanding the instructions of how to administer the drops and its storage, or just forgetfulness or the fact that they don't like to put the drops multiple times a day for 2-4 weeks, therefore they just avoid doing it.

There is a new option called "Dropless cataract surgery". This modality of treatment involves the injection of an eye compatible compound at time of cataract surgery.

The purpose of is to assess the efficacy the compound injected during routine cataract surgery and intraocular (IOL) implantation with and without a topical NSAID compared to standard prophylactic treatment that includes the topical use of Moxifloxacin, Ilevro, and Prednisolone acetate 1%.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing bilateral cataract extraction or refractive lens exchange with intraocular lens implantation.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Willing and able to administer eye drops and record the times the drops were instilled.
* Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6-15 days between surgeries.
* Potential postoperative best-corrected visual acuity of 20/30 or better

Exclusion Criteria:

* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Presence of epiretinal membrane.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* History of chronic intraocular inflammation.
* History of retinal detachment.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Previous radial keratotomy.
* Any additional ocular surgical procedures at time of cataract extraction (i.e. iStent) except corneal incisions for the correction of astigmatism.
* Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Carolina Eyecare Physicians, LLC
Locations (4):
- United States (4):
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - Ophthalmic Consultants of Long Island, Garden City, New York
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment started on December 2014 and ended in March 2016. Potential subjects were identified from the patients presenting at the clinics for eye evaluation.
Pre-assignment Details: No significant events in the study occurred after participant enrollment, but prior to randomization.
Units Other Than Participants: Eyes
Groups:
- Control: Moxifloxacin HCl 0.1%, 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  Nepafenac ophthalmic suspension 0.3% : 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Prednisolone acetate 1% will be started after surgery QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
  Moxifloxacin HCl 0.5%: Antibiotic to be used 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  Ilevro: NSAID to be used 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Prednisolone acetate 1%: Steroid to be started after surgery 1 drop QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
Period: Overall Study
Arm/Group | TriMoxiVanc | TriMoxiVanc + Ilevro | Control
Started | 29; 29 Eyes | 30; 30 Eyes | 59; 59 Eyes
Completed | 29; 29 Eyes | 26; 26 Eyes | 55; 55 Eyes
Not Completed | 0; 0 Eyes | 4; 4 Eyes | 4; 4 Eyes
Not completed — Adverse Event | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- TriMoxiVanc One Eye + Control Fellow Eye: Subject's eyes were randomized to either TriMoxiVan or Control group.
  TriMoxiVanc group:
  Triamcinolone acetonide 15 mg / ml with moxifloxacin 1 mg/ml, vancomycin 10 mg/ml used as an injection delivered into the vitreous cavity using a transzonular approach at the end of the uneventful phacoemulsification procedure after IOL implantation before removal of the OVD.
  Control group:
  Moxifloxacin HCl 0.5%: 1 drop, QID for 3 days prior to surgery and continued for 2 weeks after surgery and then discontinued.
  Ilevro (Nepafenac ophthalmic suspension 0.3%): 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Prednisolone acetate 1%: Started after surgery 1 drop QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
- TriMoxiVanc + Ilevro One Eye + Control Fellow Eye: Subject's eyes were randomized to either TriMoxiVan + Ilevro or Control group.
  TriMoxiVan + Ilevro group:
  Nepafenac ophthalmic suspension 0.3% started 3 days prior to surgery QD and continued QD for 4 weeks after surgery. The compounded Tri-Moxy-Vanco (triamcinolone acetonide 15 mg / ml with moxifloxacin 1 mg/ml, vancomycin 10 mg/ml ) injected into the vitreous cavity using a transzonular approach after IOL implantation before removal of the OVD.
  Control group:
  Moxifloxacin HCl 0.5%: 1 drop, QID for 3 days prior to surgery and continued for 2 weeks after surgery and then discontinued.
  Ilevro (Nepafenac ophthalmic suspension 0.3%): 1 drop QD starting 3 days before surgery and QD for 4 weeks after surgery.
  Prednisolone acetate 1%: Started after surgery 1 drop QID for 2 weeks, tapered to BID for 2 weeks, and then discontinued.
- Total: Total of all reporting groups
Arm/Group | TriMoxiVanc One Eye + Control Fellow Eye | TriMoxiVanc + Ilevro One Eye + Control Fellow Eye | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (7.5) | 69.3 (6.8) | 68.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Preoperative Exam) in Macular Thickness
Description: Macula is the area in the retina that is responsible for the best central vision. Changes in its thickness may occur after cataract surgery due to the normal inflammatory process that occurs postoperatively but it returns to preoperative values unless there is an underlying disease.
Time Frame: Month 1.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | TriMoxiVanc | TriMoxiVanc + Ilevro | Control
Number analyzed (Participants) | 29 | 26 | 55
Microns | 12.34 (13.05) | 10.96 (11.55) | 9.84 (15.84)

2. Secondary Outcome: Change From Baseline (Preoperative Exam) in Pachymetry (Corneal Thickness)
Description: Cornea is the clear part of the front of the eye. Normal corneal thickness is in average 0.540 mm. The corneal thickness is measured with a handheld device called pachymeter.
  An increase in corneal thickness may indicate corneal edema (swelling of the cornea) that could be seen after ocular surgery.
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | TriMoxiVanc | TriMoxiVanc + Ilevro | Control
Number analyzed (Participants) | 29 | 26 | 55
Microns | 14.44 (13.95) | 5.94 (14.07) | 4.47 (15.63)

3. Secondary Outcome: Change From Baseline (Preoperative Exam) in Intraocular Pressure (IOP)
Description: Intraocular pressure refers to the pressure inside the eye. It is measured in mmHg using a device called a tonometer. The mean IOP is 15.5 mmHg. Raised IOP after cataract surgery is common and in most cases it is transient and benign.
Time Frame: Month 1.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TriMoxiVanc | TriMoxiVanc + Ilevro | Control
Number analyzed (Participants) | 29 | 26 | 55
mmHg | -0.5 (2.8) | -1.03 (3.3) | -1.1 (3.0)

ADVERSE EVENTS:
Time Frame: In average, adverse event data was collected for 6 weeks from the time the Informed consent was signed until patient exited the study.
Description: Adverse events were classified as related to study treatment or not related. All reported adverse events were considered not related to study treatment.
Arm/Group | TriMoxiVanc | TriMoxiVanc + Ilevro | Control
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/55
Other Adverse Events (participants affected / at risk) | 3/29 | 1/26 | 5/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TriMoxiVanc (N=29) | TriMoxiVanc + Ilevro (N=26) | Control (N=55)
Dry eyes (Eye disorders) | 1 | 0 | 1
Rebound inflammation (Eye disorders) | 0 | 1 | 2
Allergic conjuctivitis (Eye disorders) | 0 | 0 | 1
Posterior vitreous detachments (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No